CLINICAL TRIAL: NCT05027607
Title: Long-term Outcome After Bascom's Pit-pick Procedure for Pilonidal Sinus Disease: a Cohort Study
Brief Title: Long-term Outcome After Pit-pick for Simple Pilonidal Sinus Disease
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PSD - pit-pick
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2021-08

CONDITIONS: Pilonidal Sinus of Natal Cleft
Keywords: Pilonidal sinus; Pit-pick; Recurrence; Pain; Day Surgery
MeSH Terms: conditions — Pilonidal Sinus; Recurrence; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bascom's pit-pick — Pit-pick procedure of simple pilonidal sinus disease in the natal cleft in a day-surgery setting.

SUMMARY:
Single-center cohort study of long-term results after pit-pcik for pilonidal sinus disease.

DETAILED DESCRIPTION:
The standard treatment at Nordsjællands Hospital in Hillerød (NOH) has since 2007 been Bascom's pit-pick procedure (PP) for simple pilonidal sinus disease (PSD), while Bascom's cleft-lift procedure has been performed in complicated cases not suitable for PP operation, recurrences following previous excisions, including PP, and unhealed midline wounds. PP operation is a minimally invasive procedure performed using local anesthesia in day surgery or outpatient clinic with certain advantages such as quick healing, less pain and a quick return to work as well as cosmetic advantages with no change to the overall appearance and shape of the gluteal cleft. The procedure is less resource demanding requiring fewer staff members and less time spent at the hospital as well as a quick return to daily life. Short-term studies showing great results following PP operation have previously been published, but so far, no long-term results have been published regarding Danish patients. Furthermore, it has previously been stated that most recurrences happen within the first 5 years following surgery. A follow-up of at least 5 years after surgery for PSD has been proposed as the gold standard. A longer follow-up is warranted to fully understand, whether PP procedure is a fully adequate treatment with an acceptable rate of recurrence and patient satisfaction or whether it only delays the time before the patients eventually undergo a final treatment.

The study is based on data of patients in a local pilonidal database. The patients in the database have all undergone surgery for pilonidal sinus disease at NOH during the period of 2007 to 2014. Data in the database has been collected prospectively up to one year following surgery and subsequently supplemented with data collected by questionnaire and telephone interviews for the period from one year follow-up and until the date of long-term follow-up. Study data were collected and managed using REDCap electronic data capture tools hosted at NOH.

Patients receive a REDCap survey per e-mail to a personal digital mailbox or are asked to participate in a telephone interview to fill out a standardized questionnaire. Patients without a personal digital mailbox receive the questionnaire by regular mail. The survey is sent out twice with a four-week interval. Only patients who do not fill out the questionnaire the first time, receive the survey a second time as a reminder. Telephone interviews are only conducted, if patients do not reply to the questionnaire received digitally or as a physical copy. The questionnaire includes questions regarding demographic characteristics, lifestyle, complications, recurrence and new interventions, pain, and cosmetic satisfaction. Medical records are reviewed to verify answers from the questionnaire if consent by the patient is given through the survey or during the telephone interview. Patients experiencing symptoms of recurrence, are offered an assessment at the hospital.

The surgical intervention: the patient is placed in a prone position and the natal cleft is kept open using tape straps. Local analgesia is administered around the midline pits and at the site of the planned lateral incision using lidocaine 5 mg/ml with adrenaline 5 µg/ml. Occasionally the procedure was performed under general anesthesia. All midline pits are identified and excised using a scalpel removing hairs and infected granulation tissue. To drain the sinus, a lateral incision is made about 1-2 cm from the midline on the most appropriate side and through this incision underlying sinuses are either curetted or excised. Additional secondary pits are removed as part of the lateral incision. Midline wounds and separately excised secondary pits close to the midline are closed with suture using transcutaneous polypropylene 3-0 or 4-0 madras suture, while the lateral incision is left open and covered with bandage and transparent film dressing to heal by secondary intention.

Risk of recurrence and time to complete wound healing is analyzed using competing risk analysis as well as univariate and multivariate Cox regression analyses including the following risk factors: sex, age, smoking, BMI, relevant co-morbidities, diabetes mellitus, acne, hidradenitis, previous interventions, preoperative abscess, number of primary and secondary pits, number of lateral incisions and postoperative complications. Remaining outcomes are analyzed as categorical variables using descriptive data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing pit-pick at Nordsjællands Hospital during the study period

Exclusion Criteria:

* Included in project investigating novel wound dressing.

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with simple pilonidal sinus disease referred to a secondary and tertiary care hospital. Prior surgery for pilonidal sinus disease included in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Treatment failure assessed by clinical assessment or by questionnaire | 10 years
  Incomplete wound healing or recurrence after complete wound healing

SECONDARY OUTCOMES:
Chronic pain related to cicatrix | 10 years
  Numerical rate scale pain score (0-10). 0 being no pain and 10 being the the worst imaginary pain
Cosmetic appearance of the cicatrix | 10 years
  Numerical rate scale score (1-5). 1 being worst, 5 the better

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, PhD, Study Chair — Department of Surgery, Copenhagen University Hospital - Nordsjaellands Hospital
Locations (1):
- Nordsjaellands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
After de-identification, individual participant data will be made available to investigators who provide a methodologically sound proposal for meta-analyses.

REFERENCES:
- [Background] Colov EP, Bertelsen CA. Short convalescence and minimal pain after out-patient Bascom's pit-pick operation. Dan Med Bull. 2011 Dec;58(12):A4348. PMID 22142576
- [Background] Serup CM, Svarre KJ, Kanstrup CTB, Kleif J, Bertelsen CA. Long-term outcome after Bascom's pit-pick procedure for pilonidal sinus disease: A cohort study. Colorectal Dis. 2023 Mar;25(3):413-419. doi: 10.1111/codi.16383. Epub 2022 Nov 13. PMID 36268754